CLINICAL TRIAL: NCT01116804
Title: Role PET Imaging in Response Assessment for Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/115
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Primary Liver Cancer
Keywords: Primary liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- inoperable liver cancer patients (Other)
  Interventions: Procedure: MRI of the liver before start of treatment; Procedure: MRI after treatment; Procedure: PET-scan before treatment start; Procedure: PET scan after treatment

INTERVENTIONS:
Procedure: MRI of the liver before start of treatment — MRI of the liver as classic work out of patients (CT-scan if MRI is contra-indicated)
Procedure: MRI after treatment — MRI of the liver after 3 - 6 months of treatment (CT-scan if MRI is contra-indicated)
Procedure: PET-scan before treatment start — PET-scan with 2 tracers is performed before treatment start
Procedure: PET scan after treatment — PET-scan with 2 tracers is repeated 4 weeks following start of treatment

SUMMARY:
Present imaging modalities for primary liver cancer (hepatocellular carcinoma or HCC) have several shortcomings. One important shortcoming is the time delay between successful treatment and radiological confirmation of this response. Often it takes several months for anatomical changes to occur and to be appreciated on morphological imaging such as CT or MRI (shrinkage of tumor, absence of contrast enhancement). Functional imaging by means of Fluor-18 deoxyglucose or Fluor-18 Choline (positron emitters, PET-scan) might be an early indicator of response. This "early" information might help to tailor treatment. For instance, if no response is induced, an early switch in therapy can be planned.

The present study investigates whether the routine PET-tracer (Fluor-18 deoxyglucose) and the experimental PET-tracer, Fluor-18 Choline help to predict response if a patient with inoperable primary liver cancer is treated (radionuclide therapy, biologicals).

ELIGIBILITY:
Inclusion Criteria :

* Male and female are eligible

  ->18years of age.No upper age limit.
* not pregnant or breastfeeding
* capable of understanding the study goals and protocol and to sign the informed consent.
* Patients are diagnosed with primary liver cancer and referred for treatment with biologicals such as Sorafenib or treatment with radionuclides.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-06-16 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of PET-imaging versus classic response assessment (MRI, CT-scam) in patients with inoperable liver cancer | 6 months after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bieke Lambert, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be